CLINICAL TRIAL: NCT06369844
Title: The Impact of 'Stop Pressure Injury' Education for Pediatric Patients on Nurses' Knowledge Level and the Probability of Pediatric Pressure Injury Occurrence
Brief Title: Pressure Injury Education Intervention for Pediatric Intensive Care Nurses: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Collaborators: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Neşe ÖZYURT, Principal İnvestigator, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1.2023-440
Record Dates: First submitted 2024-04-09; First posted 2024-04-17 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Pressure Injury Prevention
Keywords: pressure injuries; pediatric; nurses knowledge
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: The study design will be two-group and pretest-posttest design.
Who Masked: Participant, Outcomes Assessor
Masking Description: The information about which group (intervention or control) the nurses who volunteered to participate in the study would belong to was provided after the pre-test data were collected. Blinding of the researcher was not performed because the researcher conducted the educational phase of the study. The determination of the study groups was carried out randomly by a person not associated with the study using a random draw method. The statistical analysis of the study data was conducted by someone not related to the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The group that received pediatric pressure injury education
  Interventions: Other: Pressure injury education
- Control group (No Intervention): The group that did not receive pediatric pressure injury education

INTERVENTIONS:
Other: Pressure injury education — Pressure injury education will be provided to participants in the intervention group in three separate sessions covering the topics of Pressure Injury Definition and Classification, Risk Assessment, Prevention, and Care.
  Arms: Intervention group

SUMMARY:
The purpose of this observational study is to find out the impact of pressure injury education on the knowledge level of pediatric intensive care nurses and the likelihood of pediatric pressure injury occurrence. The main questions it aims to answer are:

* Does pressure injury education increase nurses knowledge level on pediatric pressure injuries?
* Does the rate of pediatric pressure injuries decrease after the education?

The researcher will compare nurses working in two separate pediatric intensive care units where similar patients are treated to see if planned education on pressure injuries affects nurses knowledge level and the rate of pediatric pressure injuries.

* Volunteer nurses participating in the study will answer pressure injury survey questions prepared by the researcher.
* Nurses in the intervention group will attend planned education sessions provided by the researcher.
* Two weeks after the completion of the education sessions, all nurses in the intervention and control groups who wish to continue participating in the study will answer the pressure injury survey questions prepared by the researcher again.

DETAILED DESCRIPTION:
Children with critical illness in intensive care units are a high-risk group for pressure injuries due to immobility and intensive medical device use (Setchell et al., 2023). The study will be conducted with nurses working in third-level pediatric intensive care units within a city hospital in Ankara. There are five pediatric intensive care units in the hospital: a 16-bed Pediatric Surgical Intensive Care Unit, a 16-bed Pediatric Cardiovascular Surgery Intensive Care Unit, a 12-bed Pediatric Intensive Care Unit, and another 12-bed Pediatric Intensive Care Unit. The number of nurses working in these intensive care units is 25, 20, 28, and 29, respectively. These 102 nurses constitute the population of the study. Firstly, the sample size was determined. G-power 3.1.9.4 analysis program was used to determine the sample size. Considering a similar study on the topic, the sample size was calculated (Karimian et al., 2020). The effect size was calculated as 1.23 in the reference study. According to this effect size, considering a 5% error rate (α) and 95% power (1-β), it was determined that there should be a total of 38 participants in the study, with 19 in the intervention group and 19 in the control group. However, assuming possible losses in the sample, the sample size was increased by 30%, resulting in 25 participants in the intervention group and 25 in the control group (n1: 25 - n2: 25). Then, considering the sample size, the pediatric intensive care units where nurses would participate in the sampling were determined. Three-month pressure injury rates of these intensive care units were obtained from the hospital's quality unit to determine these units. According to these rates, these intensive care units were ranked. The first two ranks were taken by the Pediatric Intensive Care Units. To prevent the intervention and control groups from influencing each other, one of the intensive care units was designated as the intervention group and the other as the control group. During the assignment, these intensive care units were given names A and B by a person unrelated to the study. The intervention and control groups were determined by a lottery method. There are enough nurses in the relevant intensive care units to meet the determined sample size of the study. After determining the sample size of the study, the training dates were planned. The principal investigator of the study is also the pediatric wound care nurse at the hospital. As of the planned training date, service supervisors and the researcher made two calls for pre-test participation in both the intervention and control groups. Each of the intensive care units involved in the study has 12 beds and provides care to two patients per nurse. There are 8 nurses working in shifts of 08-08 hours per day. Pre-test data collection is planned for 3 days without disrupting the operation of the intensive care units. After the pre-test data collection, a pressure injury training consisting of 3 sessions lasting 40 minutes each will be provided to the intervention group for 1 week without disrupting patient care. Although the intensive care units are on separate floors in the hospital, the nurses are separate, but the patient profiles are similar. Two weeks after the completion of the training, post-test data will be collected in a similar manner. The training will cover pressure injury definition and classification, risk factors and assessment scales for pressure injuries in children, and pressure injury prevention and care. The collected data will be analyzed and interpreted using statistical methods. Pressure injury rates in the intensive care units will be compared again after the training. The questionnaire used to measure the nurses' knowledge levels and the training were created by the principal investigator. The created training and questionnaire were sent to 10 expert doctors who are specialists in their respective fields for expert opinion. The results of the expert opinions were statistically analyzed. The Cronbach's Alpha Internal Consistency Coefficient for the questionnaire used for pre-test and post-test was calculated as a total of 0.977, which is considered highly reliable.The training content has also been found to be at a very appropriate level.

ELIGIBILITY:
Inclusion Criteria:

* Working in pediatric intensive care for more than 6 months
* Having provided pressure injury care at least once
* Voluntarily agreeing to participate in the study
* Working in intensive care where pressure injuries are commonly seen.

Exclusion Criteria:

* Having wound care certification
* Not attending all of the training sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Stop Pressure Injuries" Education Evaluation Survey | he questionnaires prepared by the researcher will be answered by both groups immediately before the training for pre-test results and two weeks after the training.
  The survey consists of subheadings: Pressure Injury Definition and Classification, Risk Assessment, Prevention, and Care. The survey comprises a total of 50 true/false statements. Participants will mark the statements as true or false. They will receive 1 point for correct answers and 0 points for incorrect answers. The total score of the survey is 50.

CONTACTS AND LOCATIONS:
Overall Officials: Neşe Özyurt, Principal Investigator — Principal Investigator
Locations (1):
- Ankara yıldırım Beyazıt Üniversitesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
NAME, SURNAME , EMAIL ADDRESS
Supporting Information: Study Protocol
Time Frame: April 2024- April 2025
URL: https://orcid.org/0000-0002-3521-3490

REFERENCES:
- [Background] undefined
- [Background] Triantafyllou C, Chorianopoulou E, Kourkouni E, Zaoutis TE, Kourlaba G. Prevalence, incidence, length of stay and cost of healthcare-acquired pressure ulcers in pediatric populations: A systematic review and meta-analysis. Int J Nurs Stud. 2021 Mar;115:103843. doi: 10.1016/j.ijnurstu.2020.103843. Epub 2020 Dec 16. PMID 33373805
- [Background] Lyren A, Brilli R, Bird M, Lashutka N, Muething S. Ohio Children's Hospitals' Solutions for Patient Safety: A Framework for Pediatric Patient Safety Improvement. J Healthc Qual. 2016 Jul-Aug;38(4):213-22. doi: 10.1111/jhq.12058. PMID 26042749
- [Background] Li Z, Lin F, Thalib L, Chaboyer W. Global prevalence and incidence of pressure injuries in hospitalised adult patients: A systematic review and meta-analysis. Int J Nurs Stud. 2020 May;105:103546. doi: 10.1016/j.ijnurstu.2020.103546. Epub 2020 Jan 31. PMID 32113142
- [Background] 1. European Pressure Ulcer Asvisory Panel, National Pressure Injury Panel, Pan Pacific Injury Alliance . (2019). Prevention and Treatment of Pressure Ulcers/İnjuries: Clinical Practice Guideline. The İnternational Guideline.